CLINICAL TRIAL: NCT02012322
Title: Coenzyme Q10 and Aging: A Planning Grant
Brief Title: UCSD Q10 and Aging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Beatrice Golomb, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: R34AG026338-01 (NIH); R34AG026338-01 (NIH)
Record Dates: First submitted 2013-12-10; First posted 2013-12-16 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Age Related Symptoms; Age Related Quality of Life Issues
Keywords: Aging; Coenzyme Q10; Q10; Quality of Life; Oxidative Stress; Mitochondrial Function; Cell Energetics; Fatigue; Ubiquinone
MeSH Terms: conditions — Fatigue | interventions — coenzyme Q10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo vs. Q10 100mg vs. Q10 300mg (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo
- Placebo vs. Q10 300mg vs. Q10 100mg (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo
- Q10 100mg vs. Placebo vs. Q10 300mg (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo
- Q10 100mg vs. Q10 300mg vs. Placebo (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo
- Q10 300mg vs. Placebo vs. Q10 100mg (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo
- Q10 300mg vs. Q10 100mg vs. Placebo (Other)
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — 100mg/day for three months
  Other Names: PharmaNord Myoquinione softgel caplets
Dietary Supplement: Coenzyme Q10 — 300mg/day for three months
  Other Names: PharmaNord Myoquinione softgel caplets
Dietary Supplement: Placebo — Three month period
  Other Names: PharmaNord matched identical softgel placebo

SUMMARY:
Goal: The investigators propose to test the feasibility of giving the supplement coenzyme Q10 (Q10) improves symptoms and subjective health in an aging population.

Rationale: Direct empirical evidence has supported benefit of Q10 to many symptoms such as fatigue, muscle pain, and cognition. In addition, Q10 has also been reported to benefit other symptoms including headaches, sleep disturbances, and breathing problems. This provides a strong rationale for testing whether Q10 will have similar benefit to these symptoms in an aging population.

Method: 44 aging subjects will participate. The design is a 9 month, randomized, double-blind, placebo-controlled crossover study. Each subject will be "crossed over" between high dose Q10 (300mg), low dose Q10 (100mg), and placebo, receiving each agent for 3 month periods. Neither subjects nor investigators will know which substance each subject is receiving in which phase. Subjects will be randomly assigned to one of six arms.

Assessments: Assessments will include feasibility of study, subjective quality of life, energy, and metabolic and lipid panels. Analyses will show whether Q10 led to improvements when compared to placebo; whether higher Q10 doses improved outcomes more than lower doses; and whether people with certain symptoms or characteristics get more benefit than people with other symptoms or characteristics.

DETAILED DESCRIPTION:
Goal: To determine feasibility of a double-blind placebo-controlled crossover study to test whether coenzyme Q10 (Q10) administration reduces symptoms and improve subjective health in an aging population.

Rationale: In a number of settings, studies have reported benefits of Q10 to fatigue, muscle pain, and cognition. Additionally Q10 defends against mechanisms that may play a role in health problems in aging populations. For these reasons, a study evaluating benefits by Q10 to symptoms and quality of life in an aging population is merited.

Subjects: 44 subjects ages 55 and older.

Design: 9 month, randomized, placebo-controlled, double-blind crossover study.

Analyses: Nonparametric and secondarily parametric analyses will compare effects of Q10 vs placebo; and of higher dose vs lower dose Q10 on primary and secondary endpoints. Possible effect modification (differential benefit) based on factors such as oxidative state and Q10 serum concentration will be explored through regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >55 years with a minimum of 40% females
* Willing to fast for 8 hrs prior to blood draw
* Must be able to complete survey instruments or assessments
* Must be independent living
* Must be community living
* Willing to defer participation in other clinical trials till after completion of study participation.
* Agree to abstain from other Q10-containing products for the duration of participation

Exclusion Criteria:

* Women who are pre-menopausal or have the capability to conceive children
* Diagnosed with HIV
* Diagnosed with cancer (except non-melanoma skin cancer)
* Diagnosed with NYHA Stage 3 or 4 congestive heart failure
* Is currently taking coumadin
* Cannot commit to continued participation for a minimum of 1 year
* Have taken Q10 including dermal preparations in the last three months
* Due to the very small number of subjects, special classes (including prisoners, institutionalized individuals, or other who may be considered vulnerable populations)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Feasibility and Acceptability (e.g., duration of study, study visits, comprehension of the quality of life questionnaires, reliability of the cognitive function measures, tolerance of study drug) | 2 years

SECONDARY OUTCOMES:
Energy (self-reported) | 2 years
Metabolic and Lipid Panel | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice A Golomb, M.D., Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD General Clinical Research Center, La Jolla, California, United States

REFERENCES:
- See also: Beatrice Golomb MD, PhD CURRICULUM VITAE — http://www.cnl.salk.edu/~bgolomb/